CLINICAL TRIAL: NCT02744690
Title: Topical vs Injection Application of Mitomycin C Trabeculectomy Trial
Brief Title: Mitomycin C Trabeculectomy Trial for Glaucoma in Ethiopia
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: The necessary ethical approvals were not obtained in a timely manner.
Sponsor: University of California, San Francisco (Other)
Collaborators: Menelik II Hospital (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 15-16075-MMC
Record Dates: First submitted 2016-02-11; First posted 2016-04-20 (Estimated); Last update posted 2023-08-01 (Actual); Status verified 2023-07

CONDITIONS: Glaucoma
Keywords: Eye Disease; Intraocular Pressure; Visual Acuity; Trabeculectomy
MeSH Terms: conditions — Glaucoma; Eye Diseases | interventions — Mitomycin

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- MMC Injection (Experimental): Intervention: At the intended surgical site and about 6mm from the limbus, 0.2ml of 0.2mg/ml of mitomycin-C (MMC) will be injected subconjunctivally before peritomy
  Interventions: Drug: Mitomycin-C (MMC)
- MMC Sponge Application (Active Comparator): Intervention: After peritomy, three half-sponges soaked in 0.2mg/ml mitomycin-C (MMC) will be placed posterior to the area of intended filtration. After 2 minutes, the sponges will be removed
  Interventions: Drug: Mitomycin-C (MMC)

INTERVENTIONS:
Drug: Mitomycin-C (MMC) — Mitomycin-C is routinely applied to the eye prior to trabeculectomy at Menelik II Hospital

SUMMARY:
This study is a randomized, double-masked trial to examine the response to trabeculectomy surgery. In this study, patients will be randomized to receive MMC via subconjunctival injection or topical sponge application.

DETAILED DESCRIPTION:
This study is a randomized, double-masked (study participants and outcome assessors) trial. During the enrollment period, patients from Menelik Hospital who are planning to have trabeculectomy surgery and who meet the study enrollment criteria will be randomized to receive mitomycin C applied topically or by injection during the surgery.At Menelik Hospital mitomycin-C (MMC) is routinely applied to the eye prior to trabeculectomy by physicians via both sponge and injection routes. The primary outcome is the patient's response to the trabeculectomy procedure, as measured by cumulative complications after a 3-month follow-up period post-operation. Secondary outcome is the change in intraocular pressure after a 3 month follow-up period. The investigators will perform subgroup analyses by stratifying the population according to skin pigmentation to determine whether pigmentation is a predictor of treatment success.

ELIGIBILITY:
Inclusion Criteria:

* Age >=40
* Planning to have a trabeculectomy

Exclusion Criteria:

* Life threatening or debilitating disease
* Inability to complete necessary exams and/or ocular disease that would preclude assessment of intraocular pressure, visual field, or optic disc
* Pseudophakic lens
* Contralateral eye already enrolled in study

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2015-03-01 (Estimated); Primary Completion 2019-03-01 (Estimated); Study Completion 2019-03-01 (Estimated)

PRIMARY OUTCOMES:
Cumulative incidence of complications | 3 months after surgery
  Comparison of the cumulative incidence of complications between the treatment groups (MMC sponge and injection application) 3 months after surgery

SECONDARY OUTCOMES:
Cumulative incidence of complications | 6 and 12 months after surgery
  Comparison of the cumulative incidence of complications between the treatment groups (sponge and injection application of MMC) 6 months and 12 months after surgery
Reduction of intraocular pressure from baseline, mmHg | 3, 6, and 12 months after surgery
  The investigators will compare the reduction of IOP from baseline between the treatment groups at 3, 6, and 12 months after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Jeremy D Keenan, MD, MPH, Principal Investigator — University of California, San Francisco
Locations (1):
- Menelik II Hospital, Addis Ababa, Ethiopia